CLINICAL TRIAL: NCT00731614
Title: Psychosocial and Visual Feedback Intervention for Phantom Limb Pain
Brief Title: Cognitive Behavior Therapy (CBT) and Mirror Training for Phantom Limb Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F6441-R; UCSD IRB 080898 (Other: UCSD IRB)
Record Dates: First submitted 2008-08-05; First posted 2008-08-11 (Estimated); Results first posted 2015-06-18 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Phantom Limb
Keywords: cognitive therapy; mirror training; nondirective therapy; veterans; amputees
MeSH Terms: conditions — Phantom Limb | interventions — Cognitive Behavioral Therapy; Palliative Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Cognitive Behavior Therapy + mirror retraining
  Interventions: Behavioral: Cognitive Behavioral Therapy and Mirror Retraining; Behavioral: Mirror retraining
- Arm 2 (Active Comparator): Supportive psychotherapy
  Interventions: Behavioral: Supportive therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy and Mirror Retraining — Cognitive Behavioral Pain Management treatment administered in 8 weeks of individual treatment, combined with training in use of a mirror device to reduce phantom limb pain.
  Arms: Arm 1
Behavioral: Supportive therapy — Non-directive, emotion focused psychotherapy to facilitate coping with pain, delivered in weekly individual sessions.
  Other Names: Non-directive therapy
  Arms: Arm 2
Behavioral: Mirror retraining — Use of a mirror to produce an illusion of the missing limb. By attending to the reflected limb while moving the existing limb, the patient provides visual feedback that helps correct changes in the neural organization of the somatosensory cortex resulting from the amputation and contributing to the phantom limb pain
  Other Names: Mirror box training
  Arms: Arm 1

SUMMARY:
The goal of this study is to test whether a combination of cognitive-behavior therapy and mirror training reduces phantom limb pain for veterans with amputations.

DETAILED DESCRIPTION:
The proposed study is a randomized controlled trial designed to test whether CBT plus mirror therapy (CBT+MT) is superior to supportive care (SC) for treatment of phantom limb pain (PLP) in amputees. The primary hypothesis is that CBT+ MT will lead to significantly greater reductions in PLP compared to SC. Secondary hypotheses will test whether CBT+MT also leads to significantly greater improvements in psychiatric symptoms, functioning, and quality of life than SC.

Eighty veterans from the San Diego VA Healthcare System (SDVAHS) will be recruited. All veterans will have a unilateral upper or lower limb amputation. All participants will complete an intake assessment prior to treatment randomization. The assessment will include measures of pain (Phantom Limb Pain Questionnaire, Descriptive Differential Scale, McGill Pain Questionnaire) psychiatric symptoms (Patient Health Questionnaire, Posttraumatic Stress disorder Checklist), psychiatric diagnosis (Mini-International Neuropsychiatric Interview) and functioning (Trinity Amputation and Prosthesis Experiences Scale, Short Form-36). Participants will then randomized to either CBT+MT or SC. Participants will complete pain and mood assessments weekly during treatment, and be retested on the full assessment battery at the end of treatment and 12 and 24 weeks posttreatment.

The CBT+MT intervention will consist of 8 individual sessions of CBT, including psychoeducation, cognitive restructuring, relaxation training, and acceptance techniques. Participants in the CBT+MT condition will also learn to use a mirror apparatus to reduce PLP, and will receive a set of mirrors to use at home. The SC treatment will consist of the therapist meeting with the patient and using listening and reflection skills to discuss the patient's pain. The SC condition will have no pain education or skills training component.

Data analyses will use a repeated-measures ANOVA approach to test whether the two conditions differ on change in the primary measure (Phantom Limb Pain Questionnaire) as well as in other pain, psychiatric symptom, functioning and quality of life measures. Exploratory analyses will test whether patient variables and amputation characteristics predict treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult (21or over)
* unilateral amputation at or above wrist or ankle
* phantom limb pain occurring at least weekly
* living within 50 miles of a recruitment site (San Diego, San Francisco, or Long Beach VAs).
* able to read and speak English

Exclusion Criteria:

* Current alcohol or drug dependence
* active psychosis
* medical problems that preclude participation
* current enrollment in behavioral pain management

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-11; Primary Completion 2011-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R. McQuaid, PhD MS BA, Principal Investigator — VA Medical Center, San Francisco
Locations (3):
- United States (3):
  - VA Medical Center, Long Beach, Long Beach, California
  - VA San Diego Healthcare System, San Diego, San Diego, California
  - VA Medical Center, San Francisco, San Francisco, California

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While 59 participant initially enrolled, 1 completed no assessments, so the overall n= 58. In addition, 4 did not complete the first week assessment session, which is why patient flow ends up listing 54 at the start rather than 58.
Groups:
- Cognitive Behavior Therapy + Mirror Retraining: Cognitive Behavioral Therapy and Mirror Retraining: Cognitive Behavioral Pain Management treatment administered in 8 weeks of individual treatment, combined with training in use of a mirror device to reduce phantom limb pain.
  Mirror retraining: Use of a mirror to produce an illusion of the missing limb. By attending to the reflected limb while moving the existing limb, the patient provides visual feedback that helps correct changes in the neural organization of the somatosensory cortex resulting from the amputation and contributing to the phantom limb pain
- Supportive Psychotherapy: Supportive therapy: Non-directive, emotion focused psychotherapy to facilitate coping with pain, delivered in weekly individual sessions.
Period: Overall Study
Arm/Group | Cognitive Behavior Therapy + Mirror Retraining | Supportive Psychotherapy
Started | 23 | 31
End of Treatment | 16 | 24
12 Weeks Posttreatment | 18 | 23
Completed | 16 | 18
Not Completed | 7 | 13

BASELINE CHARACTERISTICS:
Population: Participants are adults with a single limb amputation who report current phantom limb pain.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavior Therapy + Mirror Retraining | Supportive Psychotherapy | Total
Number analyzed (Participants) | 26 | 32 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.12 (12.85) | 54.62 (16.32) | 57.09 (14.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 23 | 30 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 18 | 21 | 39
  Unknown or Not Reported | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 18 | 23 | 41
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 26 | 32 | 58

OUTCOME MEASURES:

1. Primary Outcome: Phantom Limb Pain Questionnaire
Description: The primary outcome measure is the severity of phantom limb pain on a likert scale from 0 (no pain) to 10 (worst pain imaginable)
Time Frame: Baseline, each weekly treatment session (1-8), 12 weeks post treatment, 24 weeks posttreatment.
Population: Data analyzed for participants with complete data for all assessments using repeated measure ANOVA.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Behavior Therapy + Mirror Retraining | Supportive Psychotherapy
Number analyzed (Participants) | 9 | 14
units on a scale
  Intake Pain Severity | 6.22 (.82) | 5.71 (.66)
  Session 1 Pain Severity | 6.67 (.71) | 4.86 (.57)
  Session 2 Pain Severity | 6.00 (.88) | 4.71 (.70)
  Session 3 Pain Severity | 4.67 (.82) | 4.57 (.65)
  Session 4 Pain Severity | 4.44 (.93) | 4.79 (.75)
  Session 5 Pain Severity | 4.78 (.96) | 4.63 (.77)
  Session 6 Pain Severity | 3.33 (.87) | 3.57 (.69)
  Session 7 Pain Severity | 3.44 (.91) | 4.29 (.73)
  Session 8 Pain Severity | 4.89 (.84) | 3.64 (.68)
  12 week posttreatment Pain Severity | 4.33 (.93) | 3.93 (.75)
  24 week posttreatment Pain Severity | 4.44 (.93) | 4.00 (.74)
Statistical Analysis 1: Comparison: Cognitive Behavior Therapy + Mirror Retraining vs Supportive Psychotherapy; Conducted a repeated measures ANOVA comparing CBT+mirror retraining with Supportive Therapy across 11 time points. The primary hypothesis was a group by time interaction. Due to missing data, a total of 9 and 14 participants, respectively could be included in analyses; Test type: Superiority or Other; p = .322, Repeated Measure ANOVA

2. Secondary Outcome: Short Form-12 (SF-12)
Description: the Short Form-12 (SF-12) is a standardized self-report questionnaire that assesses mental and physical functioning. The Physical Component Summary (PCS) is scored on a scale from 0-100, with higher scores representing better reported health.
Time Frame: Baseline, end of treatment (8 weeks after baseline)
Population: While a total of 49 participants completed the trial, missing data reduced the number in each condition for some analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavior Therapy + Mirror Retraining | Supportive Psychotherapy
Number analyzed (Participants) | 21 | 28
score on a scale
  SF12 PCS baseline: number analyzed (Participants) | 18 | 23
  SF12 PCS baseline | 48.61 (11.12) | 45.58 (5.66)
  SF12 PCS 8 weeks (end of treatment): number analyzed (Participants) | 12 | 19
  SF12 PCS 8 weeks (end of treatment) | 55.47 (10.56) | 46.31 (7.48)

ADVERSE EVENTS:
Time Frame: During course of treatment (8 weekly sessions).
Arm/Group | Cognitive Behavior Therapy + Mirror Retraining | Supportive Psychotherapy
Serious Adverse Events (participants affected / at risk) | 2/23 | 3/31
Other Adverse Events (participants affected / at risk) | 1/23 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavior Therapy + Mirror Retraining (N=23) | Supportive Psychotherapy (N=31)
Admission for urinary tract infection (UTI)/urosepsis (Renal and urinary disorders) | 1 (1) | 0 — Participant had a history of chronic renal disease secondary to diabetes prior to study entry, s/p renal transplant, experienced UTI and was admitted for treatment. Symptoms were deemed unrelated to study intervention.
Peripheral arterial disease (Vascular disorders) | 1 (1) | 0 (0) — Participant withdrew from study due to deteriorating health (peripheral arterial disease). Disease progression was unrelated to study procedures.
Fall/ broken femur (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Pt fell and broke femur, requiring hospitalization and withdrawal from study. Fall was unrelated to study procedures.
Stroke (Vascular disorders) | 0 (0) | 1 (1) — Participant had stroke while driving, necessitating withdrawal from study. Stroke was unrelated to the study procedures.
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1) — Participant admitted to hospital for exacerbation of congestive heart failure due to upper respiratory infection. Hospitalization unrelated to study procedures.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavior Therapy + Mirror Retraining (N=23) | Supportive Psychotherapy (N=31)
Pain exacerbation (General disorders) | 1 (1) | 0 (0) — Participant reported increase in pain while using visual feedback for treatment of phantom limb pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes